CLINICAL TRIAL: NCT02714413
Title: Effect of D-allulose Ingestion on the Glucose and Insulin Response to a Standardized Oral Sucrose Load
Brief Title: Effect of D-allulose in Addition to Oral Sucrose Load
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IIS-Allulose-16
Record Dates: First submitted 2016-03-08; First posted 2016-03-21 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Blood Glucose
Keywords: D-allulose; Caucasian; African American
MeSH Terms: interventions — psicose; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sucrose 50g + placebo (Placebo Comparator): All the test sugars will be dissolved in 300 ml water to be consumed within 10 minutes
  Interventions: Dietary Supplement: sucrose; Other: Placebo
- Sucrose 50g + D-allulose 2.5 g (Experimental): All the test sugars will be dissolved in 300 ml water to be consumed within 10 minutes
  Interventions: Dietary Supplement: D-allulose; Dietary Supplement: sucrose
- Sucrose 50g + D-allulose 5.0 g (Experimental): All the test sugars will be dissolved in 300 ml water to be consumed within 10 minutes
  Interventions: Dietary Supplement: D-allulose; Dietary Supplement: sucrose
- Sucrose 50g + D-allulose 7.5 g (Experimental): All the test sugars will be dissolved in 300 ml water to be consumed within 10 minutes
  Interventions: Dietary Supplement: D-allulose; Dietary Supplement: sucrose
- Sucrose 50g + D-allulose10.0 g (Experimental): All the test sugars will be dissolved in 300 ml water to be consumed within 10 minutes
  Interventions: Dietary Supplement: D-allulose; Dietary Supplement: sucrose

INTERVENTIONS:
Dietary Supplement: D-allulose — Subjects will be their own controls as they will be studied sequentially for the effects of varying amounts of D-allulose given in a random order associated with standardized oral sucrose load of 50 gms. In order to limit the possibility of carry-over effect, patients will be randomized to different treatment sequences. In each sequence all four doses (2.5, 5, 7.5, and 10 gm) and placebo will be present only one time and will be administered in a different order.
  Other Names: D-psicose
  Arms: Sucrose 50g + D-allulose 2.5 g; Sucrose 50g + D-allulose 5.0 g; Sucrose 50g + D-allulose 7.5 g; Sucrose 50g + D-allulose10.0 g
Dietary Supplement: sucrose — All subjects will receive a standardized oral sucrose load of 50 gms
Other: Placebo — Subjects will be their own controls as they will be studied sequentially for the effects of varying amounts of D-allulose given in a random order associated with standardized oral sucrose load of 50 gms. In order to limit the possibility of carry-over effect, patients will be randomized to different treatment sequences. In each sequence all four doses (2.5, 5, 7.5, and 10 gm) and placebo will be present only one time and will be administered in a different order.
  Arms: Sucrose 50g + placebo

SUMMARY:
Individuals in the United States now consume a substantial proportion of their total energy as added sugars. The consumption of caloric sweeteners has been steadily increasing over the last four decades. The potential health consequences of this practice have been subject to considerable debate. In addition to weight gain, higher consumption of sugar-sweetened beverages is associated with development of metabolic syndrome and type 2 diabetes. These findings support the current dietary guidelines that encourage consumers to limit their intake of added sugars. There is a need for a sugar substitute that is safe, palatable and has favorable effects on energy metabolism and overall glucose homeostasis. One such sugar is possibly D-allulose also referred to in the literature as D-psicose. The present proposal is to address the efficacy of D-allulose in reducing postprandial blood glucose level in a random sample of Caucasian and African American population. Specifically the effect of D-allulose ingestion on the glucose and insulin response to a standardized oral glucose load will be studied.

DETAILED DESCRIPTION:
Individuals in the United States now consume a substantial proportion of their total energy as added sugars. The consumption of caloric sweeteners has been steadily increasing over the last four decades. The potential health consequences of this practice have been subject to considerable debate. In a prospective follow-up study of 43,960 African American women who gave complete dietary and weight information and were free from diabetes at baseline, the incidence of type 2 diabetes mellitus was higher with higher intake of both sugar-sweetened soft drinks and fruit drinks. Similar conclusions were drawn in a meta- analysis of 11 studies of consumption of sugar-sweetened beverages in relation to risk of metabolic syndrome and type 2 diabetes. Thus, in addition to weight gain, higher consumption of sugar-sweetened beverages is associated with development of metabolic syndrome and type 2 diabetes. These findings support the current dietary guidelines that encourage consumers to limit their intake of added sugars. There is a need for a sugar substitute that is safe, palatable and has favorable effects on energy metabolism and overall glucose homeostasis. One such sugar is possibly D-allulose also referred to in the literature as D-psicose. D-allulose is a non-calorie monosaccharide which has approximately 70% sweetness of sucrose. Early clinical trials of D-allulose demonstrating its anti-diabetic and anti-obesity effects have been carried out in Kagawa (Japan). As of to date, there are still insufficient data to confirm the efficacy of pure D-allulose in Caucasian or African American populations. The present proposal is to address the efficacy of D-allulose in reducing postprandial blood glucose level in a random sample of Caucasian and African American population. This is a single center, prospective, randomized, double-blind, placebo-controlled crossover study evaluating the efficacy of pure D-allulose in Caucasian and African American populations. Subjects will be their own controls as they will be studied sequentially for the effects of varying amounts of D-allulose given in a random order on glycemic and insulin excursions associated with standardized oral sucrose load of 50 gms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-70 years of age
* Have an HbA1C < 5.8%.
* Subjects from whom informed consent has been obtained in accordance with University of Florida Institutional Review Board regulations.

Exclusion Criteria:

* Pregnancy or lactation
* Diagnosed with diabetes mellitus
* Weight change ≥ 5 % within 3 months prior to admission to the study
* Has taken any weight loss medications within 3 months prior to admission to the study
* Immunocompromised status, including a debilitated state or malignancy
* Active liver, renal, thyroid diseases
* Frequent alcoholic consumption more than twice a week; with beer > 360 mL, alcohol > 45 mL, wine > 150 mL for female, or beer > 720 mL, whisky > 90 mL, wine > 300 mL for male each time
* Has gastrointestinal symptoms such as nausea, vomiting, loss of appetite, premature satiety, diarrhea, or chronic constipation
* Lack of ability or willingness to give informed consent
* Taken any medications than might cause weight loss or weight gain such as corticosteroid, antidepressant, antipsychotics, oral contraceptive pills < 8 weeks or change the dose of these medication with 8 week prior to admission
* People with clinical diagnosis of diabetes.
* Patients in cardiac Class II, III or IV.
* Patients who have had renal transplants or are currently receiving renal dialysis.
* Patients with the diagnosis of psychosis.
* Patients with known HIV infection.
* Patients with history of malignancy within the last one year with the exception of localized skin cancers.
* Patients with significant clinical signs or symptoms of liver disease, acute or chronic hepatitis, or aspartate transaminase (AST or SGOT) greater than three times the upper reference range limit.
* Patients with clinical signs or symptoms of drug or alcohol abuse.
* Patients with a life expectancy of less than 5 years.
* Patients with any cognitive impairment diagnosed previously
* Patients with a serum creatinine greater 1.5 mg/dl.
* Patients exhibiting serious non-compliance with prescribed diet or drug therapy.
* Patients who are currently participating or have participated in a medical, surgical, or pharmaceutical investigation in which an investigational new drug was dispensed to the patient within the last 30 days months.
* Patients with a body mass index (B.M.I.) greater than 40 kg/m2.
* Patients with a body mass index (B.M.I.) less than 20 kg/m2.
* Any situation which precludes the patient from following and completing the protocol.
* Patients with known hemoglobinopathy or chronic anemia with hemoglobin <10gm/dL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma glucose (mg/dL) | 120 minutes
  Evaluation of the efficacy of pure D-allulose on the glycemic excursion following a standard oral sucrose load.

SECONDARY OUTCOMES:
Serum insulin | 120 minutes
  Evaluation of the efficacy of pure D-allulose on the elevation of serum insulin following ingestion of a standard oral sucrose load

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franchi F, Yaranov DM, Rollini F, Rivas A, Rivas Rios J, Been L, Tani Y, Tokuda M, Iida T, Hayashi N, Angiolillo DJ, Mooradian AD. Effects of D-allulose on glucose tolerance and insulin response to a standard oral sucrose load: results of a prospective, randomized, crossover study. BMJ Open Diabetes Res Care. 2021 Feb;9(1):e001939. doi: 10.1136/bmjdrc-2020-001939. PMID 33637605